CLINICAL TRIAL: NCT03759964
Title: Ferric Carboxymaltose (Ferinject®) Administered After Cardiac Surgery: (FCAACS) Effects On Correction Of Anemia And Transfusion Rates: A Prospective Randomized Controlled Trial
Brief Title: Effects of Ferinject® on Anemia and Transfusion Rates After Cardiac Surgery
Acronym: FCAACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Collaborators: Vifor Pharma (Industry); Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Samia Madi Jebara, Professor, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEHDF 1050
Record Dates: First submitted 2018-11-25; First posted 2018-11-30 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Anemia, Iron Deficiency
Keywords: cardiac surgery; ferric carboxymaltose; anemia; transfusion
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: FCAACS will be a parallel group randomized trial, with a 2-group design and no crossover. Allocation ratio will be 1/1, in an equivalence framework.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric Carboxymaltose group (Active Comparator): Ferric carboxymaltose group will receive 1g of Ferric carboxymaltose at day 1 following cardiac surgery
  Interventions: Drug: Ferric carboxymaltose
- Placebo group (Placebo Comparator): Placebo group will receive 100 mL of IV isotonic serum saline at day 1 following cardiac surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — 1g of Ferric carboxymaltose diluted in 100 mL of IV isotonic serum saline at day 1 following surgery
  Other Names: Ferinject®
  Arms: Ferric Carboxymaltose group
Drug: Placebo — 100 mL of IV isotonic serum saline at day 1 following surgery
  Other Names: Serum saline
  Arms: Placebo group

SUMMARY:
Several studies using new forms of intravenous iron showed that it is effective in treating perioperative anemia in orthopedic and digestive surgery. Effects of ferric carboxymaltose have not been assessed in the settings of cardiac surgery.

This study will compare ferric carboxymaltose to placebo in a randomized trial design where ferric carboxymaltose / placebo will be administered in the postoperative period (Day 1) after cardiac surgery. A total sample size of 200 patients (100 per group) will be needed.

The FCAACS trial will assess the impact of administering intravenous iron (Ferric carboxymaltose) after cardiac surgery with cardiopulmonary bypass (CPB) on the:

* incidence of postoperative anemia
* incidence of postoperative transfusion
* incidence of complications related to intravenous iron

All the surgeries will be performed by the same surgical team and follow-up will be ensured by the same Cardiac Surgery Unit (CSU) team according to department's standard protocols.

Participants in the Ferric carboxymaltose group will receive 1g of Ferric carboxymaltose diluted in 100 mL of IV isotonic serum saline, whereas participants in the Placebo group will receive 100 mL of IV Placebo

DETAILED DESCRIPTION:
Anemia is very common in the perioperative of major surgery affecting about 30% of patients preoperatively and more than 80% postoperatively. Anemia is an independent risk factor of morbi-mortality.

Iron deficiency is the first cause of anemia. Physiological reserves of iron are not important, and the correction of anemia after hemorrhage is very slow. Hence, it takes 90 days to return to 80% of the basic Hb level after a blood donation of 500ml, and more than 150 days (almost 6 months), if one is deficient in iron. This is why iron is used to correct anemia that occurs after bleeding. There are two routes for iron administration: oral and intravenous.

Gastrointestinal absorption of iron is limited to 10-15 mg/d even when ingested doses are increased. This absorption is decreased in the presence of an inflammatory state, which is very common in the postoperative period.

The intravenous route allows the delivery of significantly higher doses of iron (up to 1000 mg in 1 infusion), without any limitation related to absorption. This is why it is interesting to administer it perioperatively where the expected delays are short.

There are currently new intravenous iron formulations that have two advantages: a shorter intravenous injection time and a higher maximum injectable dose per infusion. These new forms are risk-free, with no serious allergy described so far in the literature.

Several studies using new forms of intravenous iron showed that it is effective in treating perioperative anemia in orthopedic and digestive surgery. Effects of ferric carboxymaltose have not been assessed in the settings of cardiac surgery.

To assess the impact of ferric carboxymaltose in cardiac surgery, it will be compared to placebo in a randomized trial design, where ferric carboxymaltose / placebo will be administered in the postoperative period. Ferric carboxymaltose / placebo will be an add-on to the current treatment of patients in the postoperative period of cardiac surgery, the group that will be receiving placebo reflects the current management of the patients in these settings.

The FCAACS trial will assess the impact of administering intravenous iron (Ferric carboxymaltose) after cardiac surgery with cardiopulmonary bypass (CPB) on the:

* incidence of postoperative anemia
* incidence of postoperative transfusion
* incidence of complications related to intravenous iron

FCAACS will be a parallel group randomized trial, with a 2-group design and no crossover. Allocation ratio will be 1/1, in an equivalence framework. A total sample size of 200 patients (100 per group) will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for elective cardiac surgery under cardiopulmonary bypass, with no exclusion criteria, and having signed an informed consent, will be enrolled in the study.

Exclusion Criteria:

* Patients < 18 years
* Urgent surgery
* Off-pump cardiac surgery
* Redo cardiac surgery
* Preoperative anemia (Hb < 10g/l or Ht < 30%)
* Transfusion within 72h preoperatively
* Pregnancy
* History of asthma or other specific allergies
* History of allergy to iron
* Acute infection
* Hepatic insufficiency
* Renal insufficiency (creatinine Clearance < 30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Change in level of hemoglobin (g/dL) from preoperative until day 30 after surgery | Preoperative (Day -2), Day 0 [CSU admission], Day 2 [CSU discharge], Day 5 [hospital discharge], Day 30
  mean ± standard deviation, measured at 5 timepoints

SECONDARY OUTCOMES:
change in Hematocrit from preoperative until day 30 after surgery (final value) | Preoperative (Day -2), Day 0 [CSU admission], Day 2 [CSU discharge], Day 5 [hospital discharge], Day 30
  mean ± standard deviation, measured at 5 timepoints
Change in Reticulocytes count from preoperative until day 30 after surgery (final value) | Preoperative (Day -2), Day 2 [CSU discharge], Day 5 [hospital discharge], Day 30
  measured at 4 timepoints
Change in Percentage of transferrin from preoperative until day 30 after surgery (final value) | Preoperative (Day -2), Day 1 [CSU, before study drug], Day 5 [hospital discharge], Day 30
  measured at 4 timepoints
Change in Ferritin from preoperative until day 30 after surgery (final value) | Preoperative (Day -2), Day 1 [CSU, before study drug], Day 5 [hospital discharge], Day 30
  measured at 4 timepoints
Number of red cell packs transfused (final value) | Day 1, Day 5,and Day 30
  mean ± standard deviation, measured at 3 timepoints

OTHER OUTCOMES:
Total bleeding (mL) until drain removal (final value) | From Day 0 until Day 2
  mean ± standard deviation
Time to tracheal tube removal, measured in hours (final value) | From Hour 0 until Hour 6 (on average, until tracheal tube removal)
  mean ± standard deviation
Length of stay in the CSU measured in Days | From Day 0 [CSU admission] until Day 2 [on overage, CSU discharge]
  median and interquartile range
Surgical exploration for bleeding (Boolean, proportion) | From Day 0 [CSU admission] until Day 2 [on overage, CSU discharge]
  Proportion, with 95% confidence interval
Complications related to administration of Ferric carboxymaltose (proportion) | From Day 0 until Day 30
  Proportion, with 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Samia Madi-Jebara, Pr, Principal Investigator — St Joseph University Beirut
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Houry M, Tohme J, Sleilaty G, Jabbour K, Bou Gebrael W, Jebara V, Madi-Jebara S. Effects of ferric carboxymaltose on hemoglobin level after cardiac surgery: A randomized controlled trial. Anaesth Crit Care Pain Med. 2023 Feb;42(1):101171. doi: 10.1016/j.accpm.2022.101171. Epub 2022 Nov 11. PMID 36375780